CLINICAL TRIAL: NCT05211726
Title: The Effects of Added Sugar Intake on Brain Blood Flow and Hippocampal Function in Midlife Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1760500; P20GM113125 (NIH)
Record Dates: First submitted 2021-12-21; First posted 2022-01-27 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-05

CONDITIONS: Aging; Healthy Diet
Keywords: added sugars; arterial stiffness; cerebrovascular function; cognitive function

STUDY DESIGN:
Intervention Model Description: A single-blind, randomized-crossover, controlled feeding study. Participants will be provided with 10-days each of a research diet containing low sugar (LS; 5% of energy from added sugars) vs. high sugar (HS; 25% of energy from added sugars) in a random order, separated by a 2-week washout.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Added Sugar Diet (Experimental): Subjects will be provided with a diet that is low in added sugars.
  Interventions: Other: Low Added Sugar Diet
- High Added Sugar Diet (Experimental): Subjects will be provided with a diet that is high in added sugars.
  Interventions: Other: High Added Sugar Diet

INTERVENTIONS:
Other: Low Added Sugar Diet — Consumption of 10 days of a diet low in added sugars (5% of total caloric intake)
  Arms: Low Added Sugar Diet
Other: High Added Sugar Diet — Consumption of 10 days of a diet high in added sugars (25% of total caloric intake)
  Arms: High Added Sugar Diet

SUMMARY:
This study will focus on improving brain health through dietary modification of added sugars in middle aged adults (50- 64 years old). Participants will be fed two 10-day diets (one diet containing 5% of total energy from added sugars and one diet containing 25% of total energy from added sugars) and examine blood vessel function, hippocampus structure using a MRI, and memory performance.

DETAILED DESCRIPTION:
Aging is the primary risk factor for Alzheimer's disease (AD) which is the most common form of dementia and among the fastest growing causes of morbidity and mortality in the United States. The risk factors for AD emerge during midlife and are similar to cardiovascular and cerebrovascular diseases. The impact of midlife peripheral vascular changes on cardiovascular risk are worsened by poor lifestyle habits, including eating a diet that contains a lot of added sugars (defined as all caloric sweeteners added to food during processing or preparation). One effect of eating a high added sugar diet is an elevation in blood triglycerides (TGs), which impairs blood vessel function by causing inflammation; however, it is not known whether eating a lot of added sugars affects the blood vessels in the brain. The purpose of this project is to determine if there is a link between added sugar intake and brain health in midlife adults. Our hypothesis is that eating excess added sugar impairs the structure and function of an area of the brain called the hippocampus by increasing plasma TGs and systemic inflammation. To test this, we will have people eat a high and low sugar diet for 10 days each (in a random order) and test how each diet affects their blood vessel function, the structure of their hippocampus, and their memory performance. We expect to show that eating a diet that contains a lot of added sugars worsens brain health compared to a diet that contains few added sugars. The data generated from this project will help us better understand risk factors for dementia and will be used to support a future grant proposal to the National Institutes of Health aimed at lowering added sugar intake in mid-life adults and individuals with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide informed consent;
* men and postmenopausal women aged 50-64 years;
* habitual intake of added sugars ≤15% of total calories;
* systolic BP < 130 mmHg; diastolic BP < 90 mmHg;
* body mass index (BMI) <30 kg/m2 and % body fat < 25% for men and < 33% for women;
* fasting triglycerides < 200 mg/dl (< 2.3 mmol/L);
* LDL cholesterol <160 mg/dl (4.14 mmol/L);
* fasting plasma glucose <126 mg/dl (<7.0 mmol/L) and hemoglobin A1C < 6.5% at screening;
* weight stable in the prior 6 months (≤ 2 kg weight change);
* blood chemistries indicative of normal liver enzymes and renal function (estimated glomerular filtration rate using the Modification of Diet in Renal Disease (MDRD) prediction equation must be >60 ml/min/1.73 m^2).

Exclusion Criteria:

* current use of medications or supplements known to lower blood triglycerides or cholesterol (e.g., fibrates, statins, high dose niacin, high dose omega-3 supplement);
* chronic clinical diseases (e.g., coronary artery/peripheral artery/cerebrovascular diseases, heart failure, diabetes, chronic kidney disease requiring dialysis, neurological or autoimmune conditions affecting cognition (e.g. Alzheimer's disease or other form of dementia, Parkinson's disease, epilepsy, multiple sclerosis, large vessel infarct);
* major psychiatric disorder (e.g. schizophrenia, bipolar disorder);
* major depressive disorder (PHQ-9 ≥ 10);
* current or past (i.e., last 3 months) use of anti-hypertensive or other cardiovascular-acting medications known to influence vascular function and/or arterial stiffness;
* current medication use likely to affect central nervous system (CNS) functions (e.g. long active benzodiazepines);
* concussion within last 2 years and ≥ 3 lifetime concussions;
* heavy alcohol consumption (defined by the Centers for Disease Control and Prevention and United States Department of Agriculture as ≥8 drinks/week for women and ≥15 drinks/week for men).
* claustrophobia, metal implants, pacemaker or other factors affecting feasibility and/or safety of MRI scanning;
* recent major change in health status within previous 6 months (i.e., surgery, significant infection or illness);
* current smoking within the past 3 months;
* High degree of physical activity as defined by ≥ 25 leisure metabolic equivalent (MET)-hours/week, within the past 3 months.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Martens, Ph.D., Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened for inclusion in this study at the University of Delaware between January 11, 2022 - January 5, 2024. The study concluded on May 3, 2024.
Pre-assignment Details: 44 participants were consented and randomized. After baseline testing, but prior to starting the intervention, 5 participants withdrew [MRI concerns (N=3) or unable to maintain the required time commitment (N=2)]. 1 participant started the intervention, but was dropped due to a change in medication not-related to the study, thus making this participant ineligible. A total of 38 participants completed both the high and low sugar diet, with a ≥ 2-week washout in between.
Groups:
- Low Sugar, High Sugar Diet: Subjects will be provided with a diet that is low in added sugars followed by a diet that is high in added sugars.
  1. Low Added Sugar Diet: Consumption of 10 days of a diet low in added sugars (5% of total caloric intake)
  2. High Added Sugar Diet: Consumption of 10 days of a diet high in added sugars (25% of total caloric intake)
- High Sugar, Low Sugar Diet: Subjects will be provided with a diet that is high in added sugars followed by a diet that is low in added sugars.
  1. High Added Sugar Diet: Consumption of 10 days of a diet high in added sugars (25% of total caloric intake)
  2. Low Added Sugar Diet: Consumption of 10 days of a diet low in added sugars (5% of total caloric intake)
Period: Overall Study
Arm/Group | Low Sugar, High Sugar Diet | High Sugar, Low Sugar Diet
Started | 20 | 24
Completed | 18 | 20
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Sugar, High Sugar Diet | High Sugar, Low Sugar Diet | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (4) | 57 (4) | 57 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 16 | 18 | 34
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 20 | 38
Seated systolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] — Seated systolic blood pressure taken with arm at heart level after a 10-minute rest. Results are average of triplicate measurements.
  mmHg | 116 (9) | 113 (10) | 114 (10)
Seat diastolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] — Seated diastolic blood pressure taken with arm at heart level after a 10-minute rest. Results are average of triplicate measurements.
  mmHg | 70 (8) | 70 (7) | 70 (7)
Height (cm) [Mean (Standard Deviation); unit: cm] — Height measured (shoes off) on stadiometer.
  cm | 171.4 (10.6) | 170.5 (8.0) | 170.9 (9.2)
Body mass (kg) [Mean (Standard Deviation); unit: kg] — Body mass measured (shoes off) on scale.
  kg | 77.1 (16.4) | 71.2 (11.4) | 74.0 (14.2)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI calculated by using weight in kilograms (kg) divided by the square of height in meters (m2).
  kg/m^2 | 26.0 (3.4) | 24.4 (3.1) | 25.2 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Arterial Compliance (m^2 Kilopascal^-1)
Description: Change in cross-sectional area of the common carotid artery (assessed using ultrasound) per 1 mmHg increase in carotid artery blood pressure (assessed by applanation tonometry). A lower carotid artery compliance is indicative of stiffer elastic arteries.
Time Frame: Day 10 of the diet
Measure: Mean (Standard Deviation); unit: m^2 kilopascal^-1
Groups:
- High Sugar Diet: High Added Sugar Diet: Consumption of 10 days of a diet high in added sugars (25% of total caloric intake)
- Low Sugar Diet: Low Added Sugar Diet: Consumption of 10 days of a diet low in added sugars (5% of total caloric intake)
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 38 | 38
m^2 kilopascal^-1 | 0.824 (0.280) | 0.772 (0.201)

2. Primary Outcome: Cerebrovascular Reactivity (Percent Increase in Cerebral Perfusion Normalized to the Increase in PETCO2
Description: Cerebrovascular reactivity (CVR) is the relative (percent) change in total cerebral perfusion measured using pseudo-continuous arterial spin labeling per mmHg change in end-tidal carbon dioxide (ETCO2) during a brief period of hypercapnia. Hypercapnia was induced by prospective end-tidal targeting (RespirAct, Thornhill Medical) in which a target change in end-tidal CO2 of +9 millimeters of mercury (mmHg) was set. Data were only analyzed if ETCO2 changed by at least 6.5 mmHg. All data were then normalized to the absolute change in ETCO2.
Time Frame: Day 10 of the diet
Population: 5 participants did not have a CVR test with a ETCO2 changed by at least 6.5 mmHg.
  2 participants did not perform the CVR test (due to discomfortable from the mask or not adequate space in the head coil).
  MRI was quenched (not working) for 2 participant during both diets.
Measure: Mean (Standard Deviation); unit: percent increase in cerebral perfusion n
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 29 | 29
percent increase in cerebral perfusion n | 4.035 (2.486) | 6.075 (3.789)

3. Primary Outcome: Hippocampal Stiffness (kPa)
Description: Noninvasive brain imaging using Magnetic Resonance Elastography (MRE) to estimate tissue mechanical properties. Stiffness values are derived from the propagation of shear waves delivered to the head using vibration at 50 Hertz (Hz) from an acoustic driver system (Resoundant, Inc, Rochester MN) and reflects the distribution and organization of neurons, axons, and glial cells. A higher brain stiffness indicates greater tissue integrity.
  A nonlinear inversion algorithm estimated mechanical properties in the brain from acquired MRE displacement data to map shear modulus, G = G'+iG", where G' is the storage modulus and G'' is the loss modulus. From these parameters, stiffness is calculated, μ = 2*|G|^2 / (|G|+G')
Time Frame: Day 10 of the diet
Population: MRI was quenched (not working) for 2 participant during both diets. The resoundant acoustic driver system did not work for 2 participants during the Low Sugar Diet.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 36 | 34
kPa | 3.09473 (0.29062) | 3.04559 (0.30600)

4. Primary Outcome: Hippocampal Damping Ratio (Unitless Ratio)
Description: Noninvasive brain imaging using Magnetic Resonance Elastography (MRE) to estimate tissue mechanical properties. Damping Ratio is derived from the propagation of shear waves delivered to the head using vibration at 50Hz from an acoustic driver system (Resoundant, Inc, Rochester MN) and reflects the relative elasticity of the brain tissue. A lower damping ratio indicates greater tissue integrity.
  A nonlinear inversion algorithm estimated mechanical properties in the brain from acquired MRE displacement data to map shear modulus, G = G'+iG", where G' is the storage modulus and G'' is the loss modulus. From these parameters, damping ratio is calculated, ξ = G"/2*G'
Time Frame: Day 10 of the diet
Population: MRI was quenched (not working) for 2 participant during both diets. The resoundant acoustic driver system did not work for 2 participants during the LS diet.
Measure: Mean (Standard Deviation); unit: unitless ratio
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 36 | 34
unitless ratio | 0.18186 (0.02949) | 0.18794 (0.02982)

5. Primary Outcome: Revised Hopkins Verbal Learning Test (HVLT-R) Total Recall Memory
Description: The Revised Hopkins Verbal Learning Test (HVLT-R) assesses verbal learning and memory, immediate recall and delayed recall from a list of 12 words.
  Immediate recall takes place over 3 trials (out of 12 correct responses each) Total recall is the sum of trials 1-3 (out of 36 correct responses). Delayed recall takes place 20-25 minutes after trial 3 and the participant must recall the entire list of words (out of 12 correct responses).
Time Frame: Day 10 of the diet
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 38 | 38
correct responses
  Trial 1 Recall | 7.6 (1.6) | 7.8 (1.8)
  Trial 2 Recall | 9.7 (1.7) | 10.2 (1.5)
  Trial 3 Recall | 10.9 (1.3) | 11.1 (1.2)
  Total Recall | 28.2 (4.0) | 29.2 (3.9)
  Delayed Recall | 9.9 (1.9) | 10.5 (1.7)

6. Primary Outcome: Revised Brief Visuospatial Memory Test (BVMT-R) Total Recall Score
Description: The Revised Brief Visuospatial Memory Test (BVMT-R) assesses visuospatial memory and includes an immediate recall and delayed recall from images.
  Immediate recall takes place over 3 trials (out of 12 correct responses each) Total recall is the sum of trials 1-3 (out of 36 correct responses). Delayed recall takes place 20-25 minutes after trial 3 and the participant must recall or redraw all the images (out of 12 correct responses).
Time Frame: Day 10 of the diet
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 38 | 38
correct responses
  Trial 1 Recall | 5.6 (2.4) | 6.3 (2.1)
  Trial 2 Recall | 8.0 (2.3) | 8.9 (2.2)
  Trial 3 Recall | 9.3 (2.0) | 10.2 (1.8)
  Total Recall | 22.9 (6.3) | 25.2 (5.5)
  Delayed Recall | 8.9 (2.1) | 9.9 (1.8)

7. Primary Outcome: Seated Systolic Blood Pressure (mmHg)
Description: Seated systolic blood pressure taken with arm at heart level after a 10-minute rest. Results are average of triplicate measurements
Time Frame: Day 10 of diet
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 38 | 38
mmHg | 115 (10) | 111 (10)

8. Primary Outcome: Seated Diastolic Blood Pressure (mmHg)
Description: Seated diastolic blood pressure taken with arm at heart level after a 10-minute rest. Results are average of triplicate measurements
Time Frame: Day 10 of diet
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 38 | 38
mmHg | 70 (7) | 67 (7)

9. Secondary Outcome: Carotid-femoral Pulse Wave Velocity (CFPWV) (m/Seconds)
Description: Carotid-femoral pulse wave velocity (CFPWV) assessed using applanation tonometry of the carotid artery and cuff-based assessment of the femoral pulse wave (SphygmoCor XCEL). CFPWV is calculated as the distance between the carotid and femoral pulse divided by the time-delay between pulses. A higher CFPWV is indicative of stiffer elastic arteries.
Time Frame: Day 10 of the diet
Population: 1 participant did not have an accessible carotid artery via applanation tonometry for both diets
Measure: Mean (Standard Deviation); unit: m/seconds
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 37 | 37
m/seconds | 7.92 (1.00) | 7.71 (1.01)

10. Secondary Outcome: Pattern Comparison Processing Speed Test (Raw/Computed Score)
Description: National Institute of Health (NIH) Toolbox Pattern Comparison Processing Speed Test Brief, computer-based assessment of processing speed in which participants quickly determine if two visual patterns are the same or different.
  For age 50-59, raw/computed score has a mean of 41.53 and standard deviation of 19.42 based on a normative dataset (Range = 11.00 - 65.00).
  For age 60-69, raw/computed score has a mean of 39.44 and standard deviation of 16.39 based on a normative dataset (Range = 7.00 - 64.00).
  A higher score indicates a better outcome.
Time Frame: Day 10 of the diet
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 38 | 38
score on a scale | 45.50 (8.20) | 47.89 (6.29)

11. Secondary Outcome: Flanker Test (Raw/Computed Score)
Description: Brief, standardized assessment of attention and inhibitory control, which are key components of executive function.
  For age 50-59, raw/computed score has a mean of 8.21 and standard deviation of 1.73 based on a normative dataset (Range = 3.88 - 9.74).
  For age 60-69, raw/computed score has a mean of 8.16 and standard deviation of 1.60 based on a normative dataset (Range = 3.63 - 9.59).
  A higher score indicates a better outcome.
Time Frame: Day 10 of the diet
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 38 | 38
score on a scale | 8.35 (0.66) | 8.52 (0.55)

12. Secondary Outcome: Triglycerides (mg/dL)
Description: Blood biomarkers triglycerides in mg/dL
Time Frame: Day 10 of the diet
Population: 2 participants had missed blood draws on the High Sugar Diet.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High Sugar Diet | Low Sugar Diet
Number analyzed (Participants) | 36 | 38
mg/dL | 102.9 (31.0) | 91.2 (28.3)

13. Other Pre Specified Outcome: Inflammatory Cytokines (%)
Description: Biomarkers of inflammation (e.g. cytokines) from peripheral blood mononuclear cells
Time Frame: Day 10 of the diet
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Sleep Quality (%)
Description: Sleep quality will be continuously measured for 10 days using an Actiwatch.
Time Frame: Day 10 of the diet
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Oxidative Stress
Description: Blood biomarkers of oxidative stress (e.g. superoxide) using Electron Paramagnetic Resonance
Time Frame: Day 10 of the diet
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The study took place from 01/11/2022 to 05/03/2024, (e.g., 2 year, 5 months). Adverse events were monitored from baseline test to end of intervention period (completion of 10-day high and 10-day low sugar diet, including monitoring over the washout period). On average, adverse events were monitored for a total of 111 days. On average, it took 38 days to start the first diet after baseline testing. On average, the washout period was 53 days.
Description: The study contain minimal risk and all participants were considered healthy (free of disease).
  This study was a crossover design, in which participants completed the diet order as 1). low-sugar diet 2). high-sugar diet -or- 1). high-sugar diet 2). low-sugar diet.
  Adverse events are reported per diet in all participants.
Groups:
- Low Sugar Diet: Subjects will be provided with a diet that is low in added sugars followed by a diet that is high in added sugars.
  Low Added Sugar Diet: Consumption of 10 days of a diet low in added sugars (5% of total caloric intake)
- High Sugar Diet: Subjects will be provided with a diet that is high in added sugars followed by a diet that is low in added sugars.
  High Added Sugar Diet: Consumption of 10 days of a diet high in added sugars (25% of total caloric intake)
Arm/Group | Low Sugar Diet | High Sugar Diet
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT05211726/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT05211726/SAP_001.pdf
  • Informed Consent Form (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT05211726/ICF_002.pdf